CLINICAL TRIAL: NCT01086930
Title: SCIPA (Spinal Cord Injury and Physical Activity) Hands-On: Early Intensive Hand Rehabilitation After Spinal Cord Injury
Brief Title: Early Intensive Hand Rehabilitation After Spinal Cord Injury
Acronym: SCIPAHandsOn
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Austin Hospital, Melbourne Australia (Other); Hampstead Rehabilitation Centre Adelaide (Unknown); Shenton Park Rehabilitation Centre Perth (Unknown); Princess Alexandra Hospital, Brisbane, Australia (Other); Royal Rehabilitation Centre Sydney (Unknown); Prince of Wales Hospital, Sydney (Other Government); Burwood Hospital, Christchurch, New Zealand (Other)
Responsible Party: Principal Investigator, Mary Galea, Professor, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCIPA Hands-On
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): In addition to standard care participants in Group A will receive:
  • One hour of extra hand training five times per week for 8 weeks using the ReJoyce Workstation.
  The training will be supervised by a therapist and provided to the target hand. The hand exercises will be incorporated into computer games and will involve the following tasks using different manipulanda:
  * reaching
  * grasping
  * manipulating
  * pulling
  * rotating
  * releasing
  Interventions: Device: ReJoyce Workstation; Other: Standard Care
- Standard Care Group (Other): Participants in the control group will not receive any training on the instrumented workstation or electrical stimulation to the hand or upper limb. They will however continue to receive standard care as well as three 15-minute specific hand activity sessions per week specifically devoted to the practice of hand activities in a one-to-one format with a therapist (as per the treatment received by the experimental group).
  Interventions: Other: Standard Care

INTERVENTIONS:
Device: ReJoyce Workstation — The device has two parts. A muscle-stimulator garment that incorporates a wireless-triggered stimulator cuff and an earpiece, similar to a hearing aid, that sends a radio signal to the stimulator cuff. As well as a specialised workstation known as ReJoyce, which connects to a standard computer via a USB port. This work station will allow the user to play specialised computer games focusing on hand function. The stimulator system and the ReJoyce workstation were developed by Professor Arthur Prochazka, University of Alberta, Canada and has been approved by the Canadian Standards Association.
  Arms: Intervention Group
Other: Standard Care — All participants will continue to receive the same standard care for the hand and upper limb as typically provided by their rehabilitation units.

SUMMARY:
Loss of hand function is one of the most devastating consequences of tetraplegia because of the severe impact on activities of daily living (ADL) and the resultant dependency on others. This multi-centre study in 78 participants will measure whether additional hand therapy provided via an electrical stimulator glove and specialised computer workstation improves hand function in people with tetraplegia.

DETAILED DESCRIPTION:
The study is a multi-centre, assessor-blind, randomised controlled phase III trial in patients with tetraplegia (a spinal cord injury). A total of 78 participants will be randomised into two groups; 1. the experimental group and 2. the control group. The control group will receive their standard rehabilitation care, while the experimental group will receive the standard rehabilitation care plus the study treatment. The study treatment will consist of one hour of extra hand training, 5 times a week, using a specialised glove which provides electrical impulses to the patient's hand allowing them to open and close their hand. The glove will be used to play games on a specialised computer workstation which focuses on hand movement and function.

The main objective of this study is to determine if the experimental treatment is more effective than standard rehabilitation care alone in participants with tetraplegia.

Total study duration is 3 years, including an 18 month recruitment period, an 8-week treatment period followed by 6 month and 12 month follow up assessments.

The progress of the participant's therapy during the study will be assessed by a blinded assessor (the assessor will not know which group the participants are in) using standard physiotherapy and occupational therapy assessments which focus on hand function. These involve grasping and releasing different everyday objects and performing everyday tasks as well as quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they:

1. have sustained a SCI within the preceding 6 months from time of consent
2. are currently receiving inpatient rehabilitation through one of the study sites
3. will remain in hospital for 12 weeks after initial screening as part of their standard medical/rehabilitation care
4. are 16 years of age or older and able to provide informed consent
5. have a motor complete or incomplete spinal cord injury at the neurological level of C2 to T1 (as per the International Standardised Neurological Assessment for SCI)
6. can actively flex their shoulder/s to 60 degrees
7. have reduced ability to grasp using their hands
8. are able to tolerate sufficient FES to enable one hand to grasp and release
9. have the potential to benefit from FES and ReJoyce according to the judgment of the treating therapist

Exclusion Criteria:

Patients will not be included if they:

1. have any other type of neurological injury affecting the target hand (e.g. brachial plexus or peripheral nerve injuries)
2. have had recent trauma or surgery to the target hand or upper limb within the last 12 months
3. have had amputation of any digits on the target hand
4. are not able to sit out of bed each day for at least 2 hours over three consecutive days
5. have extensive fixed contractures in the upper limb of the target hand preventing use of the ReJoyce
6. have severe spasticity in the target hand or upper limb preventing use of the ReJoyce
7. are unable to attend the 6-month and 1-year follow-up assessments at their treating spinal unit
8. are likely to undergo hand surgery in the target hand in the next year
9. might experience autonomic dysreflexia and/or hypotension in response to electrical stimulation
10. have any contraindications to FES, such as cardiac pacemaker, epilepsy, forearm fracture or pregnancy
11. have intracranial metal implants
12. have impaired vision and/or are unable to view a computer screen
13. have any other serious medical condition including malignancies, psychiatric, behavioural or drug-dependency problems, which are likely to influence the participant's ability to cooperate or in the opinion of the study investigator would prevent the participant from adhering to the Protocol.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-09; Primary Completion 2012-12 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Modified Action Research Arm Test | 8 weeks and 26 weeks
  A standardized measure of unilateral hand and upper limb function

SECONDARY OUTCOMES:
Summed Upper Limb Strength of the Graded and Redefined Assessment of Strength Sensibility and Prehension | 8 weeks and 26 weeks
  Summed strength score of 10 upper limb muscles
Sensory Score on ISNCSCI | 8 weeks and 26 weeks
  Scores for light touch and pinprick tested in dermatomes of the upper limb
AsTex Sensory Test | 8 weeks and 26 weeks
  A measure of texture discrimination in the fingertips
AuSpinal Test | 8 weeks and 26 weeks
  A test of hand function
Capabilities of Upper Extremity | 8 weeks and 26 weeks
  A questionnaire about upper limb function
Assessment of Quality of Life (AQoL) | 8 weeks and 26 weeks
  A questionnaire to assess quality of life
Health Utilities Index Mark 3 | 8 weeks and 24 weeks
  A questionnaire to assess quality of life, but includes a domain on hand function
Self-care subscale of the Spinal Cord Independence Measure | 8 weeks and 24 weeks
  A questionnaire about independence in self-care
Goal Attainment Scale | 8 weeks
  An assessment of whether a participant achieved pre-set goals
Participant Perception of Treatment Effectiveness | 8 weeks
  Self resport of treatment effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Harvey, Principal Investigator — University of Sydney; Mary Galea, Principal Investigator — University of Melbourne; Sarah Dunlop, Principal Investigator — The University of Western Australia
Locations (7):
- Australia (6):
  - Spinal Unit, Prince of Wales Hospital, Randwick, New South Wales
  - Royal Rehabilitation Centre Sydney, Sydney, New South Wales
  - Queensland Spinal Cord Injury Service, Princess Alexandra Hospital, Woolloongabba, Queensland
  - South Australian Spinal Cord Injury Service, Hampstead Rehabilitation Centre, Northfield, South Australia
  - Victorian Spinal Cord Injury Service, Royal Talbot Rehabilitation Centre, Kew, Victoria
  - Sir George Bebrook Spinal Injuries Centre, Royal Perth Hospital, Shenton Park, Western Australia
- Burwood Academy, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No
Data will only be provided in aggregate. No individual data will be released, as per the ethics approval.

REFERENCES:
- [Background] Harvey LA, Dunlop SA, Churilov L, Hsueh YS, Galea MP. Early intensive hand rehabilitation after spinal cord injury ("Hands On"): a protocol for a randomised controlled trial. Trials. 2011 Jan 17;12:14. doi: 10.1186/1745-6215-12-14. PMID 21235821
- [Result] Harvey LA, Dunlop SA, Churilov L, Galea MP; Spinal Cord Injury Physical Activity (SCIPA) Hands On Trial Collaborators. Early intensive hand rehabilitation is not more effective than usual care plus one-to-one hand therapy in people with sub-acute spinal cord injury ('Hands On'): a randomised trial. J Physiother. 2016 Apr;62(2):88-95. doi: 10.1016/j.jphys.2016.02.013. Epub 2016 Mar 19. PMID 27008910
- [Derived] Harvey LA, Dunlop SA, Churilov L, Galea MP; Spinal Cord Injury Physical Activity (SCIPA) Hands On Trial Collaborators. Early intensive hand rehabilitation is not more effective than usual care plus one-to-one hand therapy in people with sub-acute spinal cord injury ('Hands On'): a randomised trial. J Physiother. 2017 Oct;63(4):197-204. doi: 10.1016/j.jphys.2017.08.005. Epub 2017 Sep 29. PMID 28970100